CLINICAL TRIAL: NCT03100799
Title: An Exploratory Clinical Study to Investigate Biomarkers of Senescence in Patients With Mild, Moderate and Severe Osteoarthritis of the Knee
Brief Title: An Exploratory Clinical Study to Investigate Biomarkers of Senescence in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UBX-OA-TNID-0001
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Senescence; Magnetic resonance imaging; Arthroscopy; Arthrocentesis; Biomarker
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroscopy; Arthrocentesis; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Single arm, exploratory non-drug, interventional biomarker study in patients with active osteoarthritis to investigate the degree of senescence-associated disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with osteoarthritis of the knee (Other): This is an exploratory non-drug, interventional biomarker study, however, there are study related procedures which are interventional such as arthroscopy, arthrocentesis and MRI assessment with infusion of a gadolinium-contrast agent.
  Interventions: Procedure: Arthroscopy; Procedure: Arthrocentesis; Diagnostic Test: MRI

INTERVENTIONS:
Procedure: Arthroscopy — Arthroscopy of the target knee
Procedure: Arthrocentesis — Arthrocentesis of the target knee and contralateral knee (if patient consents)
Diagnostic Test: MRI — MRI with and without a gadolinium-based contrast agent
  Other Names: Magnetic resonance imaging

SUMMARY:
This is an exploratory non-drug, interventional biomarker study in approximately 30 eligible patients with active osteoarthritis to investigate the degree of senescence-associated disease. Patients will provide blood and urine and undergo MRI imaging with and without gadolinium enhancement. Following imaging, arthrocentesis of both knees and an arthroscopy of the target knee will occur to obtain fluid, synovium and cartilage for analysis.

DETAILED DESCRIPTION:
This is an exploratory non-drug, interventional, hypothesis generating biomarker study. No Investigational Product will be administered in the study, however, there are study related procedures which are interventional such as arthroscopy, arthrocentesis and infusion of a gadolinium-containing contrast agent.

Consented patients who meet the selection criteria undergo MRI imaging with and without gadolinium contrast of both knees. Approximately seven days following the MRI imaging, patients undergo an arthrocentesis of both knees to obtain synovial fluid and then an arthroscopy of the target knee to obtain synovial and non-weight bearing cartilage tissues.

The patient will return to the clinic approximately seven days following the arthroscopy and arthrocentesis procedures for a routine safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed as having primary (idiopathic) femoro-tibial osteoarthritis (OA) of the knee as defined by a modified version of the American College of Rheumatology Criteria (modified clinical and laboratory criteria) for at least 6 months.
2. Kellgren-Lawrence (KL) score of grade 1 to 4 inclusive based on a standardized, semi-fixed, weight-bearing radiograph of the knee.
3. Adults of age ≥ 35 years
4. Body Mass Index less than or equal to an upper limit of 35 kg/m2
5. Patients who are able to commit the time required to attend all study visits
6. Normal clinical laboratory results with no clinically significant organ dysfunction which, in the opinion of the investigator, would preclude patient from entering the study

Exclusion Criteria:

1. Any condition, including laboratory findings and findings in the medical history or in the pre-study assessments, that, in the opinion of the Investigator constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation
2. Prior open knee surgery to the target knee including but not limited to Anterior Cruciate Ligament Repair
3. Patients who have had prior arthroscopy and intraarticular treatments for the management of osteoarthritis such as administration of hyaluronic acid or corticosteroids within the last 6 months
4. Patients with traumatic knee injury who are scheduled for arthroscopic repair procedures to either target or non-target knee
5. Patients who are deemed to be at risk of acute renal insufficiency of any severity due to hepato-renal syndrome or who are in the peri-operative liver transplant period.
6. Patients with Diabetes Mellitus.
7. Patients with renal dysfunction as defined by a Glomerular Filtration Rate <60 ml/min/1.73m2 by laboratory testing.
8. Known allergic or hypersensitivity reaction to gadolinium-based contrast agents or patients who have other contraindications for MRI
9. Patients requiring anticoagulation therapy other than low dose (81 mg or less) aspirin
10. Treatment with an unapproved investigational therapeutic agent and/or experimental therapeutic procedure on the target knee within 24 weeks prior to screening
11. Any active known or suspected systemic autoimmune disease Permitted on Study

    * vitiligo
    * residual hypothyroidism due to autoimmune condition only requiring hormone replacement
    * psoriasis not requiring systemic treatment for 2 years
    * conditions not expected to recur in the absence of an external trigger Excluded on Study
    * documented history of inflammatory bowel disease (including ulcerative colitis and Crohn's disease)
    * symptomatic autoimmune conditions (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma])
    * systemic lupus erythematosus
    * autoimmune vasculitis (e.g. Wegener's Granulomatosis)
    * patients with motor neuropathy considered of autoimmune origin (e.g. Guillain-Barré Syndrome)
12. History of previous surgery (Total or Partial Knee Replacement) on the Target knee
13. Lesions at the planned site of arthroscopy which would present a contraindication to the procedure such as open wounds or infection of the skin
14. Any known active infection, including suspicion of intra-articular infection and/or infections that may compromise the immune system such as HIV, Hepatitis B or Hepatitis C infection
15. History of sarcoma and/or history of other active malignancy within the last 5 years, except basal cell carcinoma, carcinoma in situ of the cervix and squamous cell carcinoma of the skin
16. Secondary osteoarthritis, including:

    * Joint dysplasias
    * Crystal-induced arthropathy (gout, calcium pyrophosphate deposition disease)
    * Aseptic osteonecrosis
    * Acromegaly
    * Paget's disease
    * Ehlers-Danlos Syndrome
    * Gaucher's disease
    * Stickler's syndrome
    * Joint infection
    * Hemophilia
    * Hemochromatosis
    * Neuropathic arthropathy of any cause
17. Patients with risk factors for OA of the knee (e.g.: obesity, meniscectomy) are not considered as having secondary OA and can be included in this study
18. Female patients who are pregnant. Female patients who are breast-feeding are eligible for enrollment providing the patient agrees not to breast-feed for 24 hours after receiving gadolinium for GE-MRI. Female patients of child-bearing potential must agree to utilize adequate contraceptive measures during the course of the study.
19. Patients who do not have the legal capacity or medical competency to provide consent; consent via legally authorized representative is not accepted.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Degree of synovial senescence as defined by the percentage of cells staining positive for candidate molecular markers of senescence on IHC in patients with osteoarthritis | Study Visit 3 (Day 14)
  Percentage of cells staining positive for candidate molecular markers of senescence on IHC

SECONDARY OUTCOMES:
Concentration of candidate biomarkers in serum, plasma, and urine and correlate with concentration in synovial fluid include but not limited to p16, p21, IL6 | Screening (Day 1) and Visit 3 (Day 14)
  Correlation between candidate biomarkers in serum or plasma and urine with synovial fluid biomarkers
Correlation between senescence burden in synovial tissue (percentage of cells staining positive om IHC) and synovitis (semi-quantitative scoring of synovium by gadolinium-enhanced MRI) | Visit 2 (Day 7) and Visit 3 (Day 14)
  Relationship between the synovial senescence, synovitis via biopsy samples and synovitis using gadolinium-enhanced MRI
Inter-interval variability of candidate biomarkers of senescence | Screening (Day 1) and Visit 3 (Day 14)
  Inter-interval variability of candidate biomarkers of senescence
Correlation between degree of synovitis (semi-quantitative scoring of synovium by gadolinium-enhanced MRI) with concentration of biomarkers in plasma or synovial fluid | Screening (Day 1), Visit 2 (Day 7) and Visit 3 (Day 14)
  To determine the relationship between GE-MRI-based assessment of synovium and plasma or synovial candidate biomarkers

OTHER OUTCOMES:
Correlation between senescence burden (percentage of cells staining positive on IHC) and phenotypic disease data (e.g., Kellgren Lawrence score) in patients with osteoarthritis | Screening (Day 1), Visit 2 (Day 7) and Visit 3 (Day 14)
  To explore the possible relationships between the degree of synovial senescence and other biomarkers that are identified as potentially relevant in patients with osteoarthritis
Correlation between synovitis (semi-quantitative scoring of synovium by gadolinium-enhanced MRI) and pain (WOMAC-A as derived from KOOS Knee Survey) | Screening (Day 1), Visit 2 (Day 7) and Visit 3 (Day 14)
  To explore the relationship of synovitis defined by either GE-MRI or by histologic assessment of synovial biopsy samples with WOMAC-A (as derived from the KOOS Knee Survey)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Wei, MD, Principal Investigator — The Arthritis Treatment Center
Locations (1):
- The Arthritis Treatment Center, Frederick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guermazi A, Roemer FW, Hayashi D, Crema MD, Niu J, Zhang Y, Marra MD, Katur A, Lynch JA, El-Khoury GY, Baker K, Hughes LB, Nevitt MC, Felson DT. Assessment of synovitis with contrast-enhanced MRI using a whole-joint semiquantitative scoring system in people with, or at high risk of, knee osteoarthritis: the MOST study. Ann Rheum Dis. 2011 May;70(5):805-11. doi: 10.1136/ard.2010.139618. Epub 2010 Dec 27. PMID 21187293
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Benjamini Y, Hochberg Y. Benjamini Y, Hochberg Y. Controlling the false discovery rate: a practical and powerful approach to multiple testing. J R Stat Soc B 1995;57(1):289-300.
- [Background] Kraus VB, Huebner JL, Fink C, King JB, Brown S, Vail TP, Guilak F. Urea as a passive transport marker for arthritis biomarker studies. Arthritis Rheum. 2002 Feb;46(2):420-7. doi: 10.1002/art.10124. PMID 11840444
- See also: KOOS Knee Survey — http://www.koos.nu/